### National Longitudinal Cohort of Hematological Diseases - Leukemia

(NICHE- Leukemia)

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

NCT Number: NCT04645199

National Longitudinal Cohort of Hematological Diseases- Leukemia (NICHE-Leukemia)

### Background

Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology.

### Objectives

The objectives of this study are to investigate the incidence and risk factors of leukemia and to analyze the treatment methods, prognosis and medical expenses of these patients in China.

### Subjects

Patients who were diagnosed with leukemia in the investigating hospitals from August 2, 2021.

### Method

The NICHE-Leukemia will collect basic information, diagnostic and treatment information, as well as medical expense information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

### Statistical Analysis Plan

## National Longitudinal Cohort of Hematological Diseases - Myelodysplastic Syndrome (NICHE- MDS)

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

NCT Number: NCT04645199

National Longitudinal Cohort of Hematological Diseases- Myelodysplastic Syndrome (NICHE- MDS)

### Background

Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology.

### Objectives

The objectives of this study are to investigate the incidence and risk factors of Myelodysplastic Syndrome (MDS) and to analyze the treatment methods, prognosis and medical expenses of these patients in China.

### Subjects

Patients who were diagnosed with MDS in the investigating hospitals from August 3, 2021.

### Method

The NICHE-MDS will collect basic information, diagnostic and treatment information, as well as medical expense information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

### **Statistical Analysis Plan**

## National Longitudinal Cohort of Hematological Diseases - Lymphoma

(NICHE- Lymphoma)

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

NCT Number: NCT04645199

National Longitudinal Cohort of Hematological Diseases- Lymphoma (NICHE-Lymphoma)

### Background

Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology.

### Objectives

The objectives of this study are to investigate the incidence and risk factors of Lymphoma and to analyze the treatment methods, prognosis and medical expenses of these patients in China.

### **Subjects**

Patients who were diagnosed with Lymphoma in the investigating hospitals from August 2, 2021.

### Method

The NICHE-Lymphoma will collect basic information, diagnostic and treatment information, as well as medical expense information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

### Statistical Analysis Plan

# National Longitudinal Cohort of Hematological Diseases - Bleeding Disorders (NICHE- BD)

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

NCT Number: NCT04645199

National Longitudinal Cohort of Hematological Diseases- Bleeding Disorders (NICHE-BD)

### Background

Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology.

### Objectives

The objectives of this study are to investigate the incidence and risk factors of bleeding disorders and to analyze the treatment methods, prognosis and medical expenses of these patients in China.

### **Subjects**

Patients who were diagnosed with bleeding disorders in the investigating hospitals from August 2, 2021.

### Method

The NICHE-BD will collect basic information, diagnostic and treatment information, as well as medical expense information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

### **Statistical Analysis Plan**